CLINICAL TRIAL: NCT00155324
Title: Change and Clinical Significance of Plantar Fascia Thickness After Extracorporeal Shock Wave Therapy
Brief Title: Change and Clinical Significance of Plantar Fascia Thickness After ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9361701153
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; ultrasonographic examination
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (Device)

SUMMARY:
The aim of the study is to investigate the effect of extracorporeal shock wave therapy (ESWT) on the thickness of plantar fascia measured by ultrasonographic examination among patients with chronic plantar fascitis. The change of plantar fascia thickness will be correlated with clinical improvement.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of extracorporeal shock wave therapy (ESWT) on the thickness of plantar fascia measured by ultrasonographic examination among patients with chronic plantar fascitis. Two different dosage of ESWT will be applied, and the outcome will be followed 3 and 6 months after the treatment. The change of plantar fascia thickness will be correlated with clinical improvement, including the pain improvement, foot function, and quality of life at follow up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as plantar fasciitis for at least 6 months
* refractory to other conservative treatments

Exclusion Criteria:

* Acute infection of soft tissue/bone
* Malignancy
* Epiphysiolysis in the focus
* Blood coagulation disorders
* Pregnancy
* Patients with pacemaker
* Foot deformity
* Autoimmune disorders-related arthropahy
* Sciatica
* Previous treatment with ESWT

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-10; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Thickness of plantar fascia by ultrasonographic examination at 3 & 6 months

SECONDARY OUTCOMES:
Pain (visual analogue scale) at 3 & 6 months
Foot function index at 3 & 6 months
Short Form-36 at 3 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: H W Liang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan